CLINICAL TRIAL: NCT01224925
Title: Randomized Controlled Trial of Pulp Capping Over Carious Exposures Comparing MTA With Dycal
Brief Title: RCT of Pulp Capping Over Carious Exposure in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: Norwegian Public dental health service (Unknown)
Responsible Party: Principal Investigator, Rita Kundzina, DDS,PhD (Associate professor (endodontics), University of Tromso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UiT-IKO-MTA-001
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2018-12

CONDITIONS: Carious Exposure; Human Permanent First and Second Molars; Mature Teeth; Proximal Caries; Healthy Pulp; Reversible Pulpitis
Keywords: carious exposure; pulp capping; MTA; Dycal
MeSH Terms: interventions — Dycal

STUDY DESIGN:
Intervention Model Description: Multicenter study a randomized, controlled, parallel, patient-blinded, two-arm superiority trial with a 1:1 allocation ratio
Who Masked: Participant
Masking Description: Patient -blinded
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capping over carious exposure with Dycal (Active Comparator): Total caries removal. In case of pulp exposure Direct Pulp capping with (Dycal®, Dentsply DeTrey GmbH, Konstanz, Germany)
  Interventions: Procedure: Direct pulp capping with Dycal
- Capping over carious exposure with WMTA (Experimental): Total caries removal. In case of pulp exposure Direct Pulp capping with Mineral Trioxide Aggregate White ProRoot® (WMTA) (DENTSPLY, Tulsa Dental, Tulsa, OK, USA)
  Interventions: Procedure: Direct pulp capping

INTERVENTIONS:
Procedure: Direct pulp capping with Dycal — Capping over carious exposure with Dycal. Dycal: covered with Fuji IX. After one week, part of the temporary filling was left under the permanent filling
  Other Names: (Dycal®, Dentsply DeTrey GmbH, Konstanz, Germany
  Arms: Capping over carious exposure with Dycal
Procedure: Direct pulp capping — WMTA capping over exposed pulp, wet pellet, Fuji IX. After one week, the entire temporary filling was removed,the cavity was permanently restored with a composite resin material used at the study clinic.
  Other Names: WMTA - White Mineral Trioxide Aggregate
  Arms: Capping over carious exposure with WMTA

SUMMARY:
This multicentre study was a randomized, controlled, parallel, patient-blinded, two-arm superiority trial with a 1:1 allocation ratio that followed the CONSORT guidelines.The aim of this study was to investigate whether MTA is more effective than a conventional calcium hydroxide liner (Dycal®) as a direct pulp capping material in mature molar teeth with a carious pulpal exposure.

DETAILED DESCRIPTION:
Calcium hydroxide (CH) is considered the standard material for pulp capping with good results in cases with pulpal exposure as a result of dental trauma both in animal and clinical studies. However, in carious exposures, follow-up studies of direct pulp capping performed with CH based materials have shown increasing failure rates and the outcome has been considered uncertain. Direct capping of carious exposures still remains a controversial treatment for mature teeth.

A new material, mineral trioxide aggregate (MTA) was introduced for root end filling material almost two decades ago. It is also suggested for pulp capping. MTA cement has showed good sealing ability and bio-compatibility in animal studies. Results from studies in humans corroborate the results from animal studies.

Although the overall results of pulp capping in human studies using MTA are very positive, well designed and controlled clinical studies, especially involving carious exposures on adult teeth are lacking.At the time the present study was launched, there were no RCTs comparing MTA and CH as DPC materials and the histological evaluations have primarily been based on healthy teeth, thus undermining the generalizability of the results to adult patients with carious exposures.

ELIGIBILITY:
Inclusion criteria:

* Age 18-55 years
* 1st and 2nd permanent molars
* Proximal caries to inner 1/3 of dentin (bite-wing)
* Apex closed, no periapical changes (apical radiograph)
* No periodontal pockets deeper than 4mm
* Medical history non-contributory (incl.pregnancy)
* No medication (no antibiotics during last month)
* No signs or symptoms more severe than reversible pulpitis
* Positive response to electrical pulp test(EPT) or cold test
* Written consent Inclusion requires compliance with all the criteria listed

Exclusion criteria:

* During the treatment there will be no pulpal exposure
* The bleeding of the exposed pulp cannot be controled in 10 minutes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-10-18 (Actual); Primary Completion 2015-12-10 (Actual); Study Completion 2015-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Kundzina, DDS, PhD, Principal Investigator — University of Tromso,Faculty of Health Sciences, Institute of Clinical Dentistry
Locations (4):
- Avimeda Dental Clinic, Klaipėda, Lithuania
- Norway (3):
  - Alta Dental Clinic, Alta
  - Sandessjoen Dental Clinic, Sandnessjøen
  - Tromso University Dental Clinic, Tromsø

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zander HA. Reaction of the pulp to calcium hydroxide. J Dent Res 1939;18:373-9
- [Background] Hørsted-Bindslev P, Bergenholtz G. Vital pulp therapies. In: Bergenholtz G,Hørsted-Bindslev P, Reit C. Textbook of endodontology. Blackwell Munksgaard,Oxford;2003:66-91
- [Background] Baume LJ, Holz J. Long term clinical assessment of direct pulp capping. Int Dent J. 1981 Dec;31(4):251-60. PMID 7030965
- [Background] Tronstad L. Reaction of the exposed pulp to Dycal treatment. Oral Surg Oral Med Oral Pathol. 1974 Dec;38(6):945-53. doi: 10.1016/0030-4220(74)90348-x. No abstract available. PMID 4216870
- [Background] Horsted P, Sandergaard B, Thylstrup A, El Attar K, Fejerskov O. A retrospective study of direct pulp capping with calcium hydroxide compounds. Endod Dent Traumatol. 1985 Feb;1(1):29-34. doi: 10.1111/j.1600-9657.1985.tb00555.x. No abstract available. PMID 3858095
- [Background] Barthel CR, Rosenkranz B, Leuenberg A, Roulet JF. Pulp capping of carious exposures: treatment outcome after 5 and 10 years: a retrospective study. J Endod. 2000 Sep;26(9):525-8. doi: 10.1097/00004770-200009000-00010. PMID 11199794
- [Background] Ward J. Vital pulp therapy in cariously exposed permanent teeth and its limitations. Aust Endod J. 2002 Apr;28(1):29-37. doi: 10.1111/j.1747-4477.2002.tb00364.x. PMID 12360679
- [Background] Stanley HR. Criteria for standardizing and increasing credibility of direct pulp capping studies. Am J Dent. 1998 Jan;11 Spec No:S17-34. PMID 9760878
- [Background] Torabinejad M, Watson TF, Pitt Ford TR. Sealing ability of a mineral trioxide aggregate when used as a root end filling material. J Endod. 1993 Dec;19(12):591-5. doi: 10.1016/S0099-2399(06)80271-2. PMID 8151252
- [Background] Ford TR, Torabinejad M, Abedi HR, Bakland LK, Kariyawasam SP. Using mineral trioxide aggregate as a pulp-capping material. J Am Dent Assoc. 1996 Oct;127(10):1491-4. doi: 10.14219/jada.archive.1996.0058. PMID 8908918
- [Background] Holland R, de Souza V, Nery MJ, Otoboni Filho JA, Bernabe PF, Dezan Junior E. Reaction of dogs' teeth to root canal filling with mineral trioxide aggregate or a glass ionomer sealer. J Endod. 1999 Nov;25(11):728-30. doi: 10.1016/s0099-2399(99)80118-6. PMID 10726538
- [Background] Tziafas D, Pantelidou O, Alvanou A, Belibasakis G, Papadimitriou S. The dentinogenic effect of mineral trioxide aggregate (MTA) in short-term capping experiments. Int Endod J. 2002 Mar;35(3):245-54. doi: 10.1046/j.1365-2591.2002.00471.x. PMID 11985676
- [Background] Asgary S, Parirokh M, Eghbal MJ, Ghoddusi J, Eskandarizadeh A. SEM evaluation of neodentinal bridging after direct pulp protection with mineral trioxide aggregate. Aust Endod J. 2006 Apr;32(1):26-30. doi: 10.1111/j.1747-4477.2006.00004.x. PMID 16603042
- [Background] Salako N, Joseph B, Ritwik P, Salonen J, John P, Junaid TA. Comparison of bioactive glass, mineral trioxide aggregate, ferric sulfate, and formocresol as pulpotomy agents in rat molar. Dent Traumatol. 2003 Dec;19(6):314-20. doi: 10.1046/j.1600-9657.2003.00204.x. PMID 15022999
- [Background] Farsi N, Alamoudi N, Balto K, Al Mushayt A. Clinical assessment of mineral trioxide aggregate (MTA) as direct pulp capping in young permanent teeth. J Clin Pediatr Dent. 2006 Winter;31(2):72-6. doi: 10.17796/jcpd.31.2.n462281458372u64. PMID 17315797
- [Background] Aeinehchi M, Eslami B, Ghanbariha M, Saffar AS. Mineral trioxide aggregate (MTA) and calcium hydroxide as pulp-capping agents in human teeth: a preliminary report. Int Endod J. 2003 Mar;36(3):225-31. doi: 10.1046/j.1365-2591.2003.00652.x. PMID 12657149
- [Background] Caicedo R, Abbott PV, Alongi DJ, Alarcon MY. Clinical, radiographic and histological analysis of the effects of mineral trioxide aggregate used in direct pulp capping and pulpotomies of primary teeth. Aust Dent J. 2006 Dec;51(4):297-305. doi: 10.1111/j.1834-7819.2006.tb00447.x. PMID 17256303
- [Background] Chacko V, Kurikose S. Human pulpal response to mineral trioxide aggregate (MTA): a histologic study. J Clin Pediatr Dent. 2006 Spring;30(3):203-9. doi: 10.17796/jcpd.30.3.38h13g5p84651652. PMID 16683667
- [Background] Iwamoto CE, Adachi E, Pameijer CH, Barnes D, Romberg EE, Jefferies S. Clinical and histological evaluation of white ProRoot MTA in direct pulp capping. Am J Dent. 2006 Apr;19(2):85-90. PMID 16764130
- [Background] Nair PN, Duncan HF, Pitt Ford TR, Luder HU. Histological, ultrastructural and quantitative investigations on the response of healthy human pulps to experimental capping with mineral trioxide aggregate: a randomized controlled trial. Int Endod J. 2008 Feb;41(2):128-50. doi: 10.1111/j.1365-2591.2007.01329.x. Epub 2007 Oct 23. PMID 17956562
- [Background] Bogen G, Kim JS, Bakland LK. Direct pulp capping with mineral trioxide aggregate: an observational study. J Am Dent Assoc. 2008 Mar;139(3):305-15; quiz 305-15. doi: 10.14219/jada.archive.2008.0160. PMID 18310735
- [Background] Roberts HW, Toth JM, Berzins DW, Charlton DG. Mineral trioxide aggregate material use in endodontic treatment: a review of the literature. Dent Mater. 2008 Feb;24(2):149-64. doi: 10.1016/j.dental.2007.04.007. Epub 2007 Jun 21. PMID 17586038
- [Background] Miyashita H, Worthington HV, Qualtrough A, Plasschaert A. Pulp management for caries in adults: maintaining pulp vitality. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004484. doi: 10.1002/14651858.CD004484.pub2. PMID 17443547
- [Background] Eriksen HM, Bergdahl M, Byrkjeflot LI, Crossner CG, Widstrom E, Tillberg A. Evaluation of a dental outreach teaching programme. Eur J Dent Educ. 2011 Feb;15(1):3-7. doi: 10.1111/j.1600-0579.2010.00636.x. PMID 21226799
- [Background] Bjorndal L. Stepwise excavation may enhance pulp preservation in permanent teeth affected by dental caries. J Evid Based Dent Pract. 2011 Dec;11(4):175-7. doi: 10.1016/j.jebdp.2011.09.005. PMID 22078824
- [Derived] Kundzina R, Stangvaltaite L, Eriksen HM, Kerosuo E. Capping carious exposures in adults: a randomized controlled trial investigating mineral trioxide aggregate versus calcium hydroxide. Int Endod J. 2017 Oct;50(10):924-932. doi: 10.1111/iej.12719. Epub 2016 Nov 28. PMID 27891629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four Dental Clinics
Pre-assignment Details: Ten subjects were excluded due to a lack of pulpal exposure after the complete removal of caries before assignment to groups
Groups:
- Dycal - Calcium Hydroxide Material: Pulp capping with Dycal
  Direct pulp capping over carious exposure: Dycal: covered with Fuji IX. After one week,part of the temporary filling was left under the permanent filling
- WMTA - White Mineral Trioxide Aggregate: Pulp capping with Mineral Trioxide Aggregate
  Direct pulp capping: WMTA capping over exposed pulp, wet pellet, FujiIX. After one week, the entire temporary filling was removed the cavity was permanently restored with a composite resin material used at the study clinic
Period: Overall Study
Arm/Group | Dycal - Calcium Hydroxide Material | WMTA - White Mineral Trioxide Aggregate
Started | 37 | 33
Completed | 34 | 31
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Population: We did not recorded patients sex and gender
Groups:
- WMTA - White Mineral Trioxide Aggregate: Pulp capping with Mineral Trioxide Aggregate
  Direct pulp capping: WMTA capping over exposed pulp, wet pellet, Fuji IX. After one week, the entire temporary filling was removed,the cavity was permanently restored with a composite resin material used at the study clinic
- Total: Total of all reporting groups
Arm/Group | Dycal - Calcium Hydroxide Material | WMTA - White Mineral Trioxide Aggregate | Total
Number analyzed (Participants) | 37 | 33 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (9.9) | 30.2 (9.7) | 30.6 (9.8)
Sex/Gender, Customized [Number; unit: participants] — Gender was not recorded
  participants | 0 | 0 | 0
Tooth number Upper first molar [Number; unit: participants] | 10 | 13 | 23
Upper second molar [Number; unit: participants] | 7 | 7 | 14
Lower first molar [Number; unit: participants] | 14 | 5 | 19
Lower second molar [Number; unit: participants] | 6 | 8 | 14
Cavity type Occlusial [Number; unit: participants] | 2 | 2 | 4
Mesial-occlusial [Number; unit: participants] | 16 | 13 | 29
Distal-occlusial [Number; unit: participants] | 11 | 11 | 22
Mesial-oclusial-distal [Number; unit: participants] | 8 | 7 | 15
Caries depth 2/3 into the dentine [Number; unit: participants] | 5 | 6 | 11
Caries depth >2/3 into the dentine [Number; unit: participants] | 8 | 15 | 23
Into the pulp [Number; unit: participants] | 24 | 12 | 36
Preoperative pain [Number; unit: participants]
  Pain at baseline - yes | 18 | 16 | 34
  Pain at baseline -no | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Survival of Capped Pulps
Description: Survival was defined as a non-symptomatic tooth that responded to sensibility testing and did not exhibit any periapical changes. Follow-up included pulpal testing and periapical radiograph at 6, 12, 24, and 36 months was planned . Patients who come with delay for last checkup where included in the study.
Time Frame: 44 month
Population: Three patients were lost from follow-up in Dycal group, two patients in WMTA group. Intention to treat principle (ITT) was applied; the analysis comprised all allocated cases
Measure: Mean (95% Confidence Interval); unit: Survival days
Units Other Than Participants: Tooth
Groups:
- Dycal - Calcium Hydroxide Material: Pulp capping with Dycal
  direct pulp capping over carious exposure: Dycal: covered with Fuji IX
- WMTA - White Mineral Trioxide Aggregate: Pulp capping with Mineral Trioxide Aggregate
  Direct pulp capping: WMTA capping over exposed pulp, wet pellet, FujiIX
Arm/Group | Dycal - Calcium Hydroxide Material | WMTA - White Mineral Trioxide Aggregate
Number analyzed (Participants) | 37 | 33
Number analyzed (Tooth) | 37 | 33
Survival days | 842 [693 to 991] | 1201 [1068 to 1335]
Statistical Analysis 1: Comparison: Dycal - Calcium Hydroxide Material vs WMTA - White Mineral Trioxide Aggregate; The power calculation was based on the intention to show a 30% difference in success rates. The following parameters were used (binomial scale): type I error: 5%; expected success rate in the CH group: 55% (based on Barthel et al. 2000); minimal difference between success rates not to be overlooked: 30%; type II error: 5%. The calculations revealed the need for 64 subjects in each group. After adding 20% for eventual drop-outs, we planned to recruit 160 subjects in one year; Test type: Superiority; p < 0.01, Log Rank; Log Rank (Mantel-Cox) = 842, 95% CI 2-sided [693 to 991]
Statistical Analysis 2: Comparison: Dycal - Calcium Hydroxide Material vs WMTA - White Mineral Trioxide Aggregate; Test type: Superiority; p < 0.01, Log Rank; Log Rank (Mantel-Cox) = 1201, 95% CI 2-sided [1068 to 1335]

2. Secondary Outcome: Postoperative Pain 1 Week After Treatment.
Description: Pain existing immediately postoperatively, during the first week, and at the one-week appointment is recorded.
Time Frame: one week
Population: Postoperative pain 1 week after treatment
Measure: Number; unit: participants
Groups:
- Direct Pulp Capping With Dycal: Total caries removal. In case of pulp exposure Direct Pulp capping with (Dycal®, Dentsply DeTrey GmbH, Konstanz, Germany)
  Direct pulp capping over carious exposure with Dycal: Direct pulp capping over carious exposure with Dycal.
  Dycal: covered with Fuji IX
- Direct Pulp Capping With WMTA: Total caries removal. In case of pulp exposure Direct Pulp capping with Mineral Trioxide Aggregate White ProRoot® (WMTA) (DENTSPLY, Tulsa Dental, Tulsa, OK, USA)
  Direct pulp capping: WMTA capping over exposed pulp, wet pellet, FujiIX
Arm/Group | Direct Pulp Capping With Dycal | Direct Pulp Capping With WMTA
Number analyzed (Participants) | 37 | 33
participants | 8 | 10
Statistical Analysis 1: Comparison: Direct Pulp Capping With Dycal vs Direct Pulp Capping With WMTA; Test type: Superiority; p > 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 36 month
Groups:
- Capping Over Carious Exposure With Dycal: Direct pulp capping over carious exposure: Dycal: covered with Fuji IX
- Capping Over Carious Exposure With WMTA: Direct pulp capping: WMTA capping over exposed pulp, wet pellet, FujiIX
Arm/Group | Capping Over Carious Exposure With Dycal | Capping Over Carious Exposure With WMTA
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/33
Other Adverse Events (participants affected / at risk) | 0/37 | 0/33

LIMITATIONS AND CAVEATS:
The power calculation was not performed separately for the secondary outcome, thus the analysis was underpowered and it may hide the existing differences in the occurrence of pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes